CLINICAL TRIAL: NCT01479517
Title: A Phase II, Single-Site, Open-Label Clinical Trial To Evaluate The Efficacy And Recommended Dosing Regimen Of Kovacaine Mist Administered Unilaterally For Anesthetizing Maxillary Teeth In Healthy Dental Patients
Brief Title: Open-Label Study of Efficacy and Recommended Dose of Kovacaine Mist for Anesthetizing Maxillary Teeth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Collaborators: Rho, Inc. (Industry); Triligent International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SR 2-05
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia
Keywords: operative; dental procedure
MeSH Terms: interventions — Tetracaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kovacaine Mist 0.1 mL x 4 sprays (Experimental): Total dose: 12 mg tetracaine/0.2 mg oxymetazoline
  Interventions: Drug: Kovacaine Mist 0.1 mL x 4 sprays
- Kovacaine Mist 0.2 mL x 2 sprays (Experimental): Total dose: 12 mg tetracaine/0.2 mg oxymetazoline
  Interventions: Drug: Kovacaine Mist 0.2 mL x 2 sprays
- Kovacaine Mist, 0.2 mL x 1 spray (Experimental): Total dose: 6 mg tetracaine/0.1 mg oxymetazoline
  Interventions: Drug: Kovacaine Mist 0.2 mL x 1 spray

INTERVENTIONS:
Drug: Kovacaine Mist 0.1 mL x 4 sprays — Dose = 4 intranasal sprays of study drug delivered at 4-minute intervals.
  Other Names: Tetracaine HCl 3% and HCl 0.05%
  Arms: Kovacaine Mist 0.1 mL x 4 sprays
Drug: Kovacaine Mist 0.2 mL x 2 sprays — Dose = 2 intranasal sprays of study drug delivered at 4-minute intervals.
  Other Names: Tetracaine HCl 3% and HCl 0.05%
  Arms: Kovacaine Mist 0.2 mL x 2 sprays
Drug: Kovacaine Mist 0.2 mL x 1 spray — Dose = 1 intranasal spray of study drug
  Other Names: Tetracaine HCl 3% and HCl 0.05%
  Arms: Kovacaine Mist, 0.2 mL x 1 spray

SUMMARY:
The purpose of this study is to evaluate the efficacy of and recommended dosing regimen for unilateral administration of Kovacaine Mist in inducing pulpal anesthesia of the maxillary teeth for dental procedures.

DETAILED DESCRIPTION:
This is a Phase II single-center, open-label clinical trial with three dosing regimens, designed to determine the efficacy and optimal dose of the Kovacaine Mist intranasal delivery system for inducing pulpal anesthesia of maxillary teeth numbers 4-13 (maxillary right second premolar to maxillary left second premolar). Kovacaine will be administered intranasally on the same side of the midline as the tooth on which the procedure will be performed in three dosing cohorts [four 100 μL, two 200 μL, or one 200 μL spray(s)] of 10 subjects each. The first cohort receiving 4 sprays will be completed before initiating study of the remaining two cohorts, which will be treated using a randomized, parallel-group design. Administration: Subjects in the 4- and 2-spray cohorts will be administered the same total dose of 12 mg tetracaine HCl/0.2 mg oxymetazoline HCl. The 4-spray cohort will be treated with a sequence of four 100-μL sprays at intervals of 4 minutes. The 2-spray cohort will be treated with a sequence of two 200 μL sprays 4 minutes apart. The 1-spray cohort will be administered one 200 μL spray, a total dose of 6 mg tetracaine HCl/0.1 mg oxymetazoline HCl, which is half the dose of the 2-spray cohort. Rescue: If the study drug does not provide sufficient anesthesia to allow for completion of the dental procedure, a rescue injection of articaine will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are 18 years of age or older;
* requiring an operative restorative procedure on a single maxillary tooth with no evidence of pulpal pathology requiring local anesthesia;
* having normal lip, nose, eyelid, and cheek sensations;
* able to understand and sign the informed consent document, communicate with the investigators, and understand and comply with the requirements of the protocol;
* having patency of naris on same side of head as tooth requiring the dental procedure.

Exclusion Criteria:

* Inadequately controlled hypertension (blood pressures greater than 150/90) or untreated coronary heart disease;
* inadequately controlled thyroid disease including Hashimoto's thyroiditis and partial thyroidectomy;
* having frequent nose bleeds (10 per month);
* having received dental care requiring a local anesthetic within the last 24 hours;
* history of allergy to or intolerance of tetracaine, benzyl alcohol, benzocaine, other ester local anesthetics, or para-aminobenzoic acid (as found in PABA-containing sunscreens);
* history of allergy or hypersensitivity to articaine, oxymetazoline, epinephrine, or sulfite preservatives; history of taking a monoamine oxidase inhibitor within the past 3 weeks;
* are nursing, pregnant, suspected of being pregnant, or trying to become pregnant. (Females will be required to take a urine pregnancy test on the day of but prior to study drug administration to rule out pregnancy);
* having used any investigational drug and/or participated in any clinical research trial within 30 days of baseline
* enlarged prostate
* narrow angle glaucoma
* use of oxymetazoline or phenylephrine nasal spray or oral decongestant on the day of the study
* congenital or idiopathic methemoglobinemia
* diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Sletten, DDS, Principal Investigator — Rock Dental Clinic
Locations (1):
- Rock Dental Clinic, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kovacaine Mist 0.1 mL x 4 Sprays | Kovacaine Mist 0.2 mL x 2 Sprays | Kovacaine Mist, 0.2 mL x 1 Spray
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kovacaine Mist 0.1 mL x 4 Sprays | Kovacaine Mist 0.2 mL x 2 Sprays | Kovacaine Mist, 0.2 mL x 1 Spray | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.42) | 58.6 (9.55) | 54.0 (15.2) | 54.7 (12.53)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 6 | 7 | 20
  Male | 3 | 4 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 10 | 10 | 29
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Receiving Kovacaine Mist Who do Not Require Rescue Anesthesia During the Operative Dental Procedure
Time Frame: at 15 minutes, with +10 minute window
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist 0.1 mL x 4 Sprays | Kovacaine Mist 0.2 mL x 2 Sprays | Kovacaine Mist, 0.2 mL x 1 Spray
Number analyzed (Participants) | 10 | 10 | 10
participants | 10 | 7 | 8

2. Secondary Outcome: The Incidence of Subjects Receiving Kovacaine Mist With Changes in Systolic and Diastolic Blood Pressure Exceeding +/- 25% of Preoperative Measurements Values.
Time Frame: 60 minutes
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist 0.1 mL x 4 Sprays | Kovacaine Mist 0.2 mL x 2 Sprays | Kovacaine Mist, 0.2 mL x 1 Spray
Number analyzed (Participants) | 10 | 10 | 10
participants
  Increased systolic BP >25% | 0 | 1 | 1
  Decreased systolic BP >25% | 0 | 0 | 0
  Increased diastolic BP >25% | 0 | 0 | 0
  Decreased diastolic BP >25% | 0 | 0 | 0

3. Secondary Outcome: The Proportion of Subjects Giving a Positive Response to Evaluation Question for Subjective Numbness Assessment (SNA) After the Procedure is Completed.
Time Frame: 60 minutes
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist 0.1 mL x 4 Sprays | Kovacaine Mist 0.2 mL x 2 Sprays | Kovacaine Mist, 0.2 mL x 1 Spray
Number analyzed (Participants) | 10 | 10 | 10
participants
  Lip numb | 6 | 5 | 3
  Side of nose numb | 9 | 5 | 5
  Lower eyelid numb | 3 | 0 | 0
  Cheek numb | 6 | 2 | 1
  Abnormal sensation tapping front teeth | 10 | 8 | 5
  Abnormal sensation in roof of mouth | 10 | 6 | 7

4. Secondary Outcome: Naris Examination
Description: Number of patients with an abnormal naris examination finding.
Time Frame: 60 minutes post drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Kovacaine Mist 0.1 mL x 4 Sprays | Kovacaine Mist 0.2 mL x 2 Sprays | Kovacaine Mist, 0.2 mL x 1 Spray
Number analyzed (Participants) | 10 | 10 | 10
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours post-dosing
Arm/Group | Kovacaine Mist 0.1 mL x 4 Sprays | Kovacaine Mist 0.2 mL x 2 Sprays | Kovacaine Mist, 0.2 mL x 1 Spray
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 9/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kovacaine Mist 0.1 mL x 4 Sprays (N=10) | Kovacaine Mist 0.2 mL x 2 Sprays (N=10) | Kovacaine Mist, 0.2 mL x 1 Spray (N=10)
Lacrimation increased (Eye disorders) | 0 | 3 | 4 — (tearing or watery eyes)
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 — (sensation of difficult swallowing)
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 — (likely due to dental procedure)
Adverse drug reaction (General disorders) | 0 | 1 | 0 — (not otherwise specified)
Feeling cold (General disorders) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Application site discomfort (General disorders) | 0 | 1 | 0
Application site pain (General disorders) | 0 | 1 | 1 — (burning sensation)
Dizziness (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0 — (sensation at eyelid)
Sinus headache (Nervous system disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — (post-nasal drip)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 — (sore throat)
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 — (throat numb)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — (throat swelling)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 — (intranasal stinging or burning)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 6 — (runny nose)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Intranasal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Injection Site Anaesthesia (General disorders) | 0 | 1 | 0
Dental Discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No